CLINICAL TRIAL: NCT07322913
Title: Post-Market Clinical Follow-up Registry to Evaluate the Safety and Performance of the Intervascular Vascular Grafts and Patches in Patients Undergoing Bypass, Replacement, or Repair of Aortic, Peripheral, or Carotid Arteries
Brief Title: Intervascular Post-Market Clinical Follow-Up (PMCF) Registry
Status: Recruiting | Type: Observational
Sponsor: Intervascular (Industry)
Responsible Party: Sponsor
Other Study IDs: VV-TMF-00090
Record Dates: First submitted 2025-11-20; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Carotid Artery Diseases; Aortic Diseases; Peripheral Arterial Diseases
MeSH Terms: conditions — Carotid Artery Diseases; Aortic Diseases; Peripheral Arterial Disease | interventions — Transdermal Patch

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Peripheral Arterial Disease (PAD) Cohort
  Interventions: Device: Intergard Standard - Collagen Coated Vascular Grafts and Patches; Device: Hemashield - Collagen Coated Vascular Grafts and Patches; Device: Intergard Silver - Antimicrobial Collagen Coated Vascular Grafts and Patches; Device: Intergard Synergy - Antimicrobial Collagen Coated Vascular Grafts
- Aortic Disease Cohort
  Interventions: Device: Intergard Standard - Collagen Coated Vascular Grafts and Patches; Device: Hemashield - Collagen Coated Vascular Grafts and Patches; Device: Intergard Silver - Antimicrobial Collagen Coated Vascular Grafts and Patches; Device: Intergard Synergy - Antimicrobial Collagen Coated Vascular Grafts
- Carotid Artery Disease Cohort
  Interventions: Device: Intergard Standard - Collagen Coated Vascular Grafts and Patches; Device: Hemashield - Collagen Coated Vascular Grafts and Patches

INTERVENTIONS:
Device: Intergard Standard - Collagen Coated Vascular Grafts and Patches — Intergard Standard, Collagen coated vascular grafts and patches are made of knitted (knitted or knitted ultrathin) or woven polyester. The products are coated with a highly purified form of cross-linked bovine collagen to minimize intraoperative bleeding and eliminate the need for preclotting at the time of implant. Note that the radially supported grafts have a polypropylene supportive coil designed to resist kinking and compression of extra-anatomical vascular repair, where potential unwanted mechanical compression of the graft may occur.
Device: Hemashield - Collagen Coated Vascular Grafts and Patches — Hemashield Vascular Grafts and Patches are made of knitted or woven polyester. The products are impregnated with a highly purified bovine collagen to reduce bleeding at the time of implant and thereby eliminates the operative preclotting step.
Device: Intergard Silver - Antimicrobial Collagen Coated Vascular Grafts and Patches — Intergard Silver antimicrobial collagen coated vascular grafts are made of knitted (knitted or knitted ultrathin) or woven polyester. The Hemapatch Silver Ultrathin is a surgical patch made from knitted ultrathin polyester fabric. The products are coated with a highly purified form of cross-linked bovine collagen to minimize intraoperative bleeding and eliminate the need for preclotting at the time of implant. In addition to collagen coating, the collagen matrix of Intergard Silver vascular grafts and patches is loaded with an antimicrobial agent: silver acetate. The coating of silver is designed to inhibit the microbial colonization on the device and within tissue immediately proximate to the device in the acute post-operative phase.
  Groups: Aortic Disease Cohort; Peripheral Arterial Disease (PAD) Cohort
Device: Intergard Synergy - Antimicrobial Collagen Coated Vascular Grafts — Intergard Synergy antimicrobial collagen coated vascular grafts are made of knitted (knitted or knitted ultrathin) polyester. The products are coated with a highly purified form of cross-linked bovine collagen to minimize intraoperative bleeding and eliminate the need for preclotting at the time of implant.
  In addition to collagen coating, the collagen matrix of Intergard Synergy Antimicrobial collagen coated vascular grafts is loaded with antimicrobial agents: silver acetate and triclosan. The addition of silver acetate and triclosan on collagen coated vascular products is designed to inhibit the microbial colonization on the device and in the surrounding tissues in the acute postoperative phase.
  Groups: Aortic Disease Cohort; Peripheral Arterial Disease (PAD) Cohort

SUMMARY:
The purpose of this registry is to evaluate the long-term safety and performance of Intervascular Vascular Grafts and Patches (Intergard Standard, Hemashield, Intergard Silver, Intergard Synergy) for bypass, repair or replacement of aortic, peripheral, or carotid arteries. This registry is intended to further define the expected product lifetime of the devices and to collect data related to usefulness of the antimicrobial coatings.

ELIGIBILITY:
Inclusion Criteria:

* Willing, and able to provide legally-effective written informed consent (as required by Institutional Review Board or Ethics Committee)
* Male and female patients that have undergone bypass, replacement or repair of the peripheral arteries, aorta, or carotid artery using the Intervascular Vascular Grafts and Patches (Intergard Standard, Hemashield, Intergard Silver, Intergard Synergy)
* Were at least 18 years of age at the time of the procedure
* Available records for data collection with a minimum of 3 years (36 months) of data/follow-up.

Exclusion Criteria:

* Active infection in the region of device placement at the time of implantation of the Intergard Standard and Hemashield Vascular Graft or Patch.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An approximate 1,200 participants (400 treated for Aortic Disease, 400 treated for Peripheral Arterial Disease, and 400 treated for Carotid Artery Disease) from up to 25 sites across the United States and Europe will participate in this registry. The number of participants and sites included will ensure a representation of the overall population, specifically in vascular surgery. No mandated procedures, assessments or visits will be implemented, given the non-interventional and retrospective nature of the registry.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Peripheral Arterial Disease Cohort: Cohort: Percentage of participants meeting primary device patency | Procedure/surgery through registry completion, anticipated average of 5 years
  Primary device patency defined as freedom from device occlusion or reintervention
Aortic Disease Cohort: Percentage of participants meeting primary device patency | Procedure/surgery through registry completion, anticipated average of 5 years
  Primary device patency defined as freedom from device occlusion or reintervention
Carotid Artery Disease Cohort: Percentage of participants achieving freedom from occlusion or reintervention | Procedure/surgery through registry completion, anticipated average of 5 years
Peripheral Arterial Disease Cohort: Incidence of Major Adverse Limb Events (MALE) | Procedure/surgery through registry completion, anticipated average of 5 years
  MALE defined as major amputation or major reintervention, including placement of a new bypass graft, interposition graft, thrombectomy, or thrombolysis
Aortic Disease Cohort: Incidence of Major Adverse Event (MAE) | Procedure/surgery through registry completion, anticipated average of 5 years
  MAE defined as major bleeding or major reintervention
Devices with antimicrobial coating: Percentage of participants achieving freedom from infection | Procedure/surgery through registry completion, anticipated average of 5 years
  Freedom from infection defined as freedom from device-related infection following the procedure
Carotid Artery Disease Cohort: Incidence of Major Adverse Event (MAE) | Procedure/surgery through registry completion, anticipated average of 5 years
  MAE defined as major bleeding, or stroke

SECONDARY OUTCOMES:
All cohorts: Percentage of participants achieving technical success | Procedure/surgery through registry completion, anticipated average of 5 years
  Technical success defined as restoration of flow or repair of a vessel without any device deficiencies
All cohorts: Incidence of reported complications and events | Procedure/surgery through registry completion, anticipated average of 5 years
  Reported complications and events include device infection, registry or device-related serious incident or death
All cohorts: Incidence of infection | Procedure/surgery through 30 days
Peripheral Arterial Disease Cohort: Percentage of patients meeting primary-assisted device patency | Procedure/surgery through registry completion, anticipated average of 5 years
  Primary-assisted device patency is defined as freedom from device occlusion irrespective of whether an intervention was performed
Peripheral Arterial Disease Cohort: Percentage of patients meeting secondary device patency | Procedure/surgery through registry completion, anticipated average of 5 years
  Secondary device patency is defined as freedom from "permanent" loss of device patency determined through the last follow-up time point for each patient
Peripheral Arterial Disease Cohort: Rate of change in Rutherford Category | Procedure/surgery through registry completion, anticipated average of 5 years
Peripheral Arterial Disease Cohort: Rate of change in Ankle-Brachial Index | Procedure/surgery through registry completion, anticipated average of 5 years
Aortic Disease Cohort: Percentage of patients meeting primary-assisted device patency | Procedure/surgery through registry completion, anticipated average of 5 years
  Primary-assisted device patency is defined as freedom from device occlusion irrespective of whether an intervention was performed
Aortic Disease Cohort: Percentage of patients meeting secondary device patency | Procedure/surgery through registry completion, anticipated average of 5 years
  Secondary device patency is defined as freedom from "permanent" loss of device patency determined through the last follow-up time point for each patient

CONTACTS AND LOCATIONS:
Overall Officials: Director, Clinical Affairs, Study Director — Getinge
Locations (2):
- CHU Dijon Bourgogne, Dijon, France
- Hospital Universitario de Navarra, Pamplona, Spain

IPD SHARING:
Plan to Share IPD: No